CLINICAL TRIAL: NCT01519765
Title: Buccal Versus Vaginal Misoprostol for Third Trimester Induction of Labor: Randomized Control Trial
Brief Title: Buccal Versus Vaginal Misoprostol for Third Trimester Induction of Labor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ram Parvataneni MD, MPH, Associate Clinical Professor of Obstetrics and Gynecology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCLA IRB#11-002056
Record Dates: First submitted 2012-01-05; First posted 2012-01-27 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buccal misoprostol+placebo vaginal pill (Experimental)
  Interventions: Drug: Buccal Misoprostol
- Vaginal Misoprostol+placebo buccal pill (Active Comparator)
  Interventions: Drug: Vaginal misoprostol

INTERVENTIONS:
Drug: Buccal Misoprostol — Buccal rather than Vaginal misoprostol for induction of labor
  Other Names: Cytotec
  Arms: Buccal misoprostol+placebo vaginal pill
Drug: Vaginal misoprostol — Vaginal rather than buccal misoprostol for induction of labor
  Other Names: Cytotec
  Arms: Vaginal Misoprostol+placebo buccal pill

SUMMARY:
Approximately 22% of term pregnancies are induced. Misoprostol, a prostaglandin E1 analogue, is a widely accepted induction agent, that has been proven safe and effective for induction of labor. It stimulates both cervical ripening and uterine contractions, thus making it an ideal induction agent for unfavorable cervices. Research has examined the pharmacokinetics of different administration routes and effects on uterine contractility, side effects, and safety. Vaginal misoprostol has been shown to be superior over oral administration however patients often prefer a more tolerable route. Buccal administration has already been shown to be as effective as vaginal misoprostol for cervical ripening and induction in both first trimester and second trimester abortions. There is minimal research comparing buccal versus vaginal for third trimester induction of labor. The investigators study is a prospective, double blinded, randomized control trial comparing vaginal misoprostol and buccal misoprostol in equal dosages of 25 mcg. The investigators seek to answer the question whether buccal misoprostol is as effective as vaginal misoprostol for third trimester induction of labor.

DETAILED DESCRIPTION:
Design Overview This will be a prospective, double blind, randomized, placebo-controlled trial comparing buccal versus vaginal misoprostol in equal doses (25 mcg every 4 hours). Each participant will receive one buccal and one vaginal tablet, only one containing misoprostol. The administration will be repeated every four hours if contractions are inadequate (frequency less than every 5 minutes) until the cervix is favorable, spontaneous rupture of membranes occurs, or the patient is in active labor. Patient will be continued on intermittent fetal heart monitoring 1 hour after administration. Prior to discharge women in the study will be asked to complete a questionnaire as to their preferences of route of administration and side effects.

1. Recruitment, Consenting, and Confirming Eligibility: Women with obstetric, medical, or psychosocial indications of induction of labor at University of California, Los Angeles Ronald Reagan Medical Center will be evaluated for participation. Those who meet eligibility criteria will be invited to participate. The subject will be counseled about the study, and if interested, will undergo the consent process. Each potential subject will receive a thorough overview of the study protocol and will review the consent form with study staff. All questions will be answered. The subject will be advised that a decision not to participate in the study will not affect the quality or availability of medical services she will receive at the hospital. She will also be advised that she can stop participating in the study at any time, for any reason, and that this will not impact the services she receives. If the subject elects to participate, two copies of the consent will be signed by the subject and research staff. A signed consent, along with a copy of the Experimental Subjects Bill of Rights, will be given to the subject. The other consent will be filed in a locked file cabinet.

   A general medical and gynecological history and physical will be done as is standard of care. Routine obstetric labs and any other medically indicated labs will be sent as is standard of care. Patients will undergo a non-stress test and uterine contraction monitoring prior to induction of labor. Obstetrical ultrasound will be reviewed or performed if indicated per the physician. Assessment of the cervix and Bishop score, pelvis, fetal size, and presentation will be performed. An unfavorable cervix is defined as Bishop score of 6 or less (ACOG). Women with ruptured membranes will not be able to participate. Gestational age will be determined on the basis of last menstrual period, confirmed by earliest ultrasound, or a corrected estimated date of confinement by the earliest ultrasound.
2. Misoprostol Administration/ Evaluation: The subject will be randomized to either of two groups. Each participant will receive both a vaginal and buccal tablet, with one tablet containing misoprostol. Subjects will be instructed by a nurse regarding buccal placement and to swallow any residue remaining after 20 minutes.

   Intravaginal administration of pill will be performed by a resident Physician or midwife. The subject will remain recumbent for at least 30 minutes. The subject will undergo fetal heart rate (FHR) and uterine contraction monitoring for at least 1 hour after misoprostol administration. The subject may undergo further FHR and uterine contraction monitoring per physician discretion. If the subject does not have adequate uterine contractions (uterine contraction occurring at least every 5 minutes), the same dosage and route of administration regimen will be repeated to 6 maximum dosage (maximum of 150mcg). Cervical assessment of Bishop score will be performed with each treatment during vaginal administration.

   Treatment will continue until spontaneous rupture of membranes, active labor, or favorable cervix (Bishop >6). Augmentation of labor using pitocin may start after 4 hours of last misoprostol dose according to routine protocol. Amniotomy may be performed at the discretion of the managing obstetrician. If labor is not achieved after receiving 150mcg of misoprostol, it will be categorized as a failed induction. At this time, the subject may be offered oxytocin induction, foley bulb mechanical dilation, or cesarean section, according to the fetal and participant condition. Terbutaline 0.25mg subcutaneous may be given for tachysystole (5 uterine contractions in 10 minutes) with FHR changes or FHR category II-III changes (minimal variability, prolonged deceleration, repetitive variables, sinusoidal pattern, repetitive late deceleration) that are not responsive to resuscitative measures ( oxygen supplementation, side positioning, intravenous fluids) according to physician's discretion.
3. Follow up: A short survey questionnaire assessing gastrointestinal side effects, experiences, and preferences of route of administration will be given prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate / consent in a placebo-controlled trial
* Age 18 and older
* Pregnancy between 34 and 42 years of gestation
* Admitted for labor induction because of either medical, obstetric, or psychosocial indications
* Live singleton fetus
* Bishop score less than or equal to six
* Cephalic presentation
* Reactive non-stress test or Negative contraction test

Exclusion Criteria:

* Premature rupture of membranes
* Multiparity > 5
* Contraindication to vaginal or labor delivery
* Suspected placental abruption
* Significant hepatic, renal or cardiac disease
* Known hypersensitivity to misoprostol or prostaglandin analogue
* Recent prostaglandin administration for induction of labor
* Multifetal pregnancy
* Macrosomia > 4500g estimated fetal weight by ultrasound or leopold

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ram Parvataneni, MD, Principal Investigator — Associate Clinical Professor
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- See also: UCLA Department of Obstetrics and Gynecology — http://obgyn.ucla.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Buccal Misoprostol: Participants received misoprostol 25 mcg via buccal route and placebo pill via vaginal route.
  The same regimen was then repeated every four hours according to protocol.
- Vaginal Misoprostol: Participants received misoprostol 25 mcg via vaginal route and placebo pill via buccal route. This same regimen was repeated every four hours according to protocol.
Period: Overall Study
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Started | 37 | 36
Completed | 34 | 34
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 73 participants were recruited to the study. 5 participants were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (6.3) | 30 (6.51) | 29.3 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
Gestational age [Median (Full Range); unit: weeks] | 40.2 [35.8 to 41.8] | 40.8 [35.3 to 42.3] | 40.5 [35.3 to 42.3]
Bishop score [Median (Full Range); unit: scores on a scale] — The Bishop score grades patients who would be most likely to achieve a successful induction. If the Bishop score is 6 or less the chances of having a vaginal delivery are low. The score is calculated by taking the sum of five subscales of the vaginal examination: dilation, effacement, station, position, and consistency. Subscale score range 0 (worse outcome) to 3 ( better outcome). Total score range= 0 (worse outcome) to 13 (better outcome)
  The Bishop score is assessed upon admission. Patients were included in this study if their Bishop score was 6 or less.
  scores on a scale | 3 [1 to 6] | 3 [0 to 3.1] | 3 [0 to 6]
Parity [Number; unit: participants] — 1. Multiparous is defined as parity of 1 or greater
  2. Nulliparous is defined as parity of 0
  participants
    Multiparous | 9 | 9 | 18
    Nulliparous | 25 | 25 | 50
Induction indication [Number; unit: participants] — 1. Postdates included gestational ages greater than 40 weeks.
  2. Hypertensive disorder included chronic hypertension, gestational hypertension, preeclampsia, eclampsia, and HELLP.
  3. Diabetes included all gestational diabetics, Type I, and Type II diabetics.
  4. Oligohydramnios was defined as amniotic fluid index (AFI) less than 5 or deep vertical pocket less than 2.
  participants
    Post dates | 15 | 16 | 31
    Hypertensive disorder | 4 | 7 | 11
    Diabetes | 3 | 2 | 5
    Elective | 7 | 3 | 10
    Oligohydramnios | 1 | 3 | 4
    Cholestasis | 2 | 2 | 4
    Other | 2 | 1 | 3
Fetal anomaly [Number; unit: participants] — Fetal anomaly was defined as any known congenital malformation diagnosed prior to admission.
  participants | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Delivery Within 24 Hours of Labor Induction
Description: Percentage of participants able to achieve vaginal delivery within 24 hours of labor induction.
Time Frame: Within 24 hours of labor induction
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Buccal Misoprostol: Participants received misoprostol 25 mcg via buccal route and placebo pill via vaginal route.
  This same regimen was then repeated every four hours according to protocol.
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 14.7 [2.6 to 26.8] | 23.5 [9.1 to 38]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; A consecutive sample will be used as women are recruited. Based on an 80% power and an alpha of 0.05, a sample size of 103 subjects in each arm is required to detect a 20% difference between deliveries within 24hrs between the two treatment arms. An effect size of 20% was selected as this is thought to be a clinically significant difference. This is based on the Wing study showing 50% delivery within 24 hrs with vaginal misoprostol; Test type: Superiority or Other; p = 0.1611, Fisher Exact

2. Secondary Outcome: Time to Vaginal Delivery
Description: Time from start of induction to vaginal delivery was computed in participants who achieved vaginal delivery.
Time Frame: Start of induction until vaginal delivery
Population: Participants who achieved vaginal delivery were included in the analysis
Measure: Median (Full Range); unit: hours
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 20 | 24
hours | 33.3 [18.1 to 55.1] | 26.5 [3.7 to 44.9]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.018, t-test, 2 sided

3. Secondary Outcome: Time to Delivery
Description: Time from induction to delivery. All participants were included.
Time Frame: Until delivery
Measure: Median (Full Range); unit: hours
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
hours | 34.1 [18 to 36.7] | 27.5 [3.7 to 68.8]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.0623, Kruskal-Wallis

4. Secondary Outcome: Time to Active Labor
Description: Time from induction to active labor. Active labor defined as 4 cm and above. P-value computed by Kruskal-Wallis test.
Time Frame: Until active labor
Measure: Median (Full Range); unit: hours
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
hours | 22.1 [0 to 47] | 19.4 [2.3 to 40.5]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.1141, Kruskal-Wallis

5. Secondary Outcome: Rates of Vaginal Delivery
Description: Percentage of participants who delivered vaginally
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 58.8 [42.3 to 75.4] | 70.6 [55.3 to 85.9]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.4469, Fisher Exact

6. Secondary Outcome: Cesarean Delivery Rate
Description: Percentage of participants who underwent a cesarean delivery was computed. P-value was computed using Fisher's exact test.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 41.2 [24.4 to 58] | 29.4 [13.9 to 45]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.4469, Fisher Exact

7. Secondary Outcome: Number of Misoprostol Doses
Description: Number of misoprostol 25 mcg doses used during induction of labor.
Time Frame: Until delivery
Measure: Median (Full Range); unit: doses
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
doses | 2 [1 to 6] | 2 [1 to 5]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.093, Kruskal-Wallis

8. Secondary Outcome: Arrest of Dilation
Description: Percentage of participants who presented with arrest of dilation. Arrest of dilation was determined by the delivering physician.
  P-value was computed using Fisher exact test.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 29.4 [13.9 to 45] | 14.7 [2.6 to 26.8]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.2417, Fisher Exact

9. Secondary Outcome: Failed Induction of Labor
Description: Percentage of participants who were determined as a failed induction of labor. Failed induction was defined as no cervical change despite 24 hours of pitocin or 12 hours of pitocin after rupture of membranes.
  P value was computed by Fisher exact test.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 1, Fisher Exact

10. Secondary Outcome: Pitocin
Description: Percentage of patients that used pitocin during labor. P-values were computed using Fisher exact test.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 97.1 [91.3 to 102.8] | 82.4 [69.3 to 95.4]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.1054, Fisher Exact

11. Secondary Outcome: Foley Bulb
Description: Percentage of participants that required foley bulb use.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 38.2 [21.7 to 54.8] | 41.2 [24.4 to 58]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.8043, Fisher Exact

12. Secondary Outcome: Artificial Rupture of Membranes (AROM)
Description: Percentage of participants that required AROM
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 64.7 [48.4 to 81] | 67.6 [51.7 to 83.6]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.797, Fisher Exact

13. Secondary Outcome: Abnormal Fetal Heart Tracing (FHT)
Description: Feta heart tracing was reviewed for every participant until 4 hours from last misoprostol dose.
  Percentage of participants who presented with abnormal fetal heart tracing was computed.
  Abnormal fetal heart tracing was defined as category 2 and 3 fetal heart tracing according to standard criteria.
  Abnormal fetal heart tracing included any of the following tachycardia, bradycardia without absent variability, minimal variability, absent variability with or without recurrent decelerations, marked variability, prolonged deceleration and recurrent late deceleration, sinusoidal pattern.
  P values were computed by Fisher exact test.
Time Frame: Until 4 hours of last misoprostol dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 15.2 [2.7 to 27.6] | 20.6 [6.8 to 34.4]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.751, Fisher Exact

14. Secondary Outcome: Tachysystole With Abnormal FHT
Description: Feta heart tracing was reviewed for every participant until 4 hours from last misoprostol dose.
  Percentage of participants who presented with tachysystole and abnormal fetal heart tracing was computed.
  Abnormal fetal heart tracing was defined as category 2 and above. Tachysystole was defined as more than 5 uterine contractions within 10 minutes. P values were computed by Fisher exact test.
Time Frame: Until 4 hours after last misoprostol dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 5.9 [0 to 13.9] | 8.8 [0 to 18.5]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.6244, Fisher Exact

15. Secondary Outcome: Tachysystole
Description: Fetal heart tracing was reviewed until 4 hours after last misoprostol dose. Percentage of participant with tachysystole were computed. Tachysystole was defined as more than five uterine contractions in 10 minutes. P value was computed using Fisher exact test
Time Frame: Until 4 hours after last misoprostol dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 26.5 [11.4 to 41.5] | 32.4 [16.4 to 48.3]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.7906, Fisher Exact

16. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: Percentage of participants whose baby was admitted to NICU was computed from time to delivery to time of hospital discharge.
  P-value was computed using Fisher Exact test.
Time Frame: Until discharge from hospital
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 20.6 [6.8 to 34.4] | 11.8 [0.8 to 22.8]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.5118, Fisher Exact

17. Secondary Outcome: Meconium
Description: Percentage of participants who developed meconium was computed. Presence of meconium was evaluated by the delivering physician. P-value was computed using Fisher exact test.
Time Frame: Until delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 23.5 [9.1 to 38] | 23.5 [9.1 to 38]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 1, Fisher Exact

18. Secondary Outcome: Chorioamnionitis
Description: Percentage of participants affected with chorioamnionitis
Time Frame: Until 48 hours after delivery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 34 | 34
percentage of participants | 17.6 [4.6 to 30.7] | 14.7 [2.6 to 26.8]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.741, Fisher Exact

19. Secondary Outcome: APGARS
Description: Median (APGAR) score at 5 minutes after delivery. APGAR: Appearance, Pulse, Grimace, Activity, Respiration Apgar scale is determine by evaluating a newborn on 5 categories on a scale from 0 to 2, then summing up the five values.
  Score range is 0 to 10. Score above 7 are generally normal. Score below 3 may indicated poor status.
Time Frame: 5 minutes after delivery
Measure: Median (Full Range); unit: score
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 32 | 34
score | 9 [6 to 9] | 9 [7 to 9]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.579, Kruskal-Wallis

20. Secondary Outcome: Patient Satisfaction With Buccal Versus Vaginal Misoprostol Administration.
Description: All patients were given a patient satisfaction survey. Patients were asked to use a Likert scale to rate their experience on the following:
  Likert sub-scale: 1 to 5
  1=Not at all/ Never to 5= Very Much/ Always
  1. Nausea and vomiting 1=better outcome 5=worse outcome
  2. effectiveness of misoprostol 1=worse outcome 5=better outcome
  3. concerns of misoprostol 1=better outcome 5=worse outcome
  4. overall labor experience 1=worse outcome 5=better outcome Patients will be followed for the duration of their labor(usually up to 72hrs). The satisfaction survey will be conducted after delivery but will evaluate side effects that they recollect in labor.
Time Frame: Until 72 hours after delivery
Population: Patient surveys were requested from all participants however incomplete patient survey collection was obtained.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 21 | 25
units on a scale
  Nausea/ Vomiting | 1 [1 to 4] | 1 [1 to 3]
  Effectiveness | 4 [1 to 5] | 4 [1 to 5]
  Patient Concern | 2 [1 to 4] | 1 [1 to 5]
  Labor satisfaction | 4 [1 to 5] | 4 [1 to 5]
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Score for Nausea and vomiting; Test type: Superiority or Other; p = .8062, Kruskal-Wallis
Statistical Analysis 2: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Effectiveness; Test type: Superiority or Other; p = 0.1505, Kruskal-Wallis
Statistical Analysis 3: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Patient concern; Test type: Superiority or Other; p = 0.1223, Kruskal-Wallis
Statistical Analysis 4: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Labor satisfaction; Test type: Superiority or Other; p = 0.5380, Kruskal-Wallis — Patient satisfaction

21. Secondary Outcome: Patient Preference
Description: All patients were given a patient satisfaction survey after delivery. They were asked to select their preference for misoprostol intervention type: buccal, vaginal, or either.
Time Frame: Until 72 hours after delivery
Population: All participants were given the survey however incomplete collection was obtained.
Measure: Number; unit: participants
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 21 | 25
participants
  Buccal | 19 | 18
  Vaginal | 1 | 3
  Either | 1 | 4
Statistical Analysis 1: Comparison: Buccal Misoprostol vs Vaginal Misoprostol; Test type: Superiority or Other; p = 0.2868, Chi-squared — This is the overall p value of all rows

ADVERSE EVENTS:
Arm/Group | Buccal Misoprostol | Vaginal Misoprostol
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

LIMITATIONS AND CAVEATS:
Limitations to the trial were termination of study due to poor recruitment, leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No